CLINICAL TRIAL: NCT01157676
Title: Open Vs Robotic-Assisted Radical Cystectomy: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dipen J Parekh, MD, Chairman of Urology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120408; R01CA155388 (NIH); 36911 (Other: Investigator-Assigned ID)
Record Dates: First submitted 2010-06-30; First posted 2010-07-07 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Bladder Cancer Requiring Cystectomy
Keywords: open cystectomy; robotic assisted radical cystectomy; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Non inferiority phase 3 randomized clinical trial comparing robotic to open radical cystectomy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open cystectomy (Active Comparator): Open cystectomy performed using an incision made just above or at the level of umbilicus to the pubic symphysis.
  Interventions: Procedure: Open radical cystectomy
- Robotic assisted radical cystectomy (Active Comparator): Robotic assisted Radical Cystectomy (RARC) is accomplished by a robot assisted laparoscopic approach.
  Interventions: Procedure: Robotic assisted radical cystectomy; Device: DaVinci robot

INTERVENTIONS:
Procedure: Open radical cystectomy — Standard of care removal of urinary bladder.
  Arms: Open cystectomy
Procedure: Robotic assisted radical cystectomy — Standard of care removal of urinary bladder using DaVinci robot.
  Arms: Robotic assisted radical cystectomy
Device: DaVinci robot — DaVinci robotic surgical system.
  Arms: Robotic assisted radical cystectomy

SUMMARY:
This is a multi-institutional, randomized trial evaluating oncologic, perioperative, and functional outcomes following two standard care procedures for radical cystectomy. The participants will have one of the standard care procedures as part of their care. The two procedures that will be followed are open radical cystectomy and robotic assisted radical cystectomy (RARC). Open cystectomy is considered to be the more traditional approach. While newer, RARC is considered to be equivalent to open surgery when it is performed by a trained robotics surgeon. The reported complication rates of RARC appear comparable to open surgery. This means there is no significant difference in the risk between the two standard procedures. However, despite these potential advantages, true comparison between the open and robotic technique with regards to long term cancer related and functional outcomes has not been accomplished because previous studies did not compare patients of equal health status. The researchers hope to learn whether or not patients undergoing RARC recover more quickly than or at the same rate as patients undergoing an open radical cystectomy while having non inferior cancer related outcomes. This study is funded by the National Institutes of Health (NIH).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have biopsy proven bladder cancer. Official pathology report reviewed at the participating institution is required.
2. Bladder cancer must be clinical stage T1-T4, N0-1, M0. (AJCC 7th edition) or refractory cis (carcinoma in situ).

Exclusion Criteria:

1. Inability to give informed consent.
2. Prior major abdominal and pelvic open surgical procedures that would preclude a safe robotic approach, as determined by the treating surgeon.
3. At the discretion of the treating surgeon, any pre-existing condition such as severe chronic obstructive pulmonary disease that precludes a safe initiation or maintenance of pneumoperitoneum over a prolonged period of time and during surgery.
4. Age <18 or >99 years.
5. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dipen J Parekh, MD, Principal Investigator — University of Miami
Locations (16):
- United States (16):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California, Irvine Medical Center (UC Irvine), Orange, California
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at San Antonio, Medical Arts & Research Center, San Antonio, Texas
  - University of Virginia Health Science Center, Department of Urology, Charlottesville, Virginia
  - Cancer Research and Biostatistics (Data Management and Statistical Office), Seattle, Washington

REFERENCES:
- [Derived] Venkatramani V, Reis IM, Gonzalgo ML, Swain S, Svatek RS, Parekh DJ. Comparison of Complication and Readmission Rates Between Robot-Assisted and Open Radical Cystectomy: Results From the Randomized RAZOR Clinical Trial. J Urol. 2025 Jun;213(6):684-692. doi: 10.1097/JU.0000000000004497. Epub 2025 Mar 13. PMID 40080805
- [Derived] Venkatramani V, Reis IM, Gonzalgo ML, Castle EP, Woods ME, Svatek RS, Weizer AZ, Konety BR, Tollefson M, Krupski TL, Smith ND, Shabsigh A, Barocas DA, Quek ML, Dash A, Parekh DJ. Comparison of Robot-Assisted and Open Radical Cystectomy in Recovery of Patient-Reported and Performance-Related Measures of Independence: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2148329. doi: 10.1001/jamanetworkopen.2021.48329. PMID 35171260
- [Derived] Parekh DJ, Reis IM, Castle EP, Gonzalgo ML, Woods ME, Svatek RS, Weizer AZ, Konety BR, Tollefson M, Krupski TL, Smith ND, Shabsigh A, Barocas DA, Quek ML, Dash A, Kibel AS, Shemanski L, Pruthi RS, Montgomery JS, Weight CJ, Sharp DS, Chang SS, Cookson MS, Gupta GN, Gorbonos A, Uchio EM, Skinner E, Venkatramani V, Soodana-Prakash N, Kendrick K, Smith JA Jr, Thompson IM. Robot-assisted radical cystectomy versus open radical cystectomy in patients with bladder cancer (RAZOR): an open-label, randomised, phase 3, non-inferiority trial. Lancet. 2018 Jun 23;391(10139):2525-2536. doi: 10.1016/S0140-6736(18)30996-6. PMID 29976469

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Radical Cystectomy: Standard of care treatment
- Robotic Assisted Radical Cystectomy: Standard of care treatment using DaVinci robot
Period: Enrollment
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Started | 174 | 176
Completed | 174 | 176
Not Completed | 0 | 0
Period: Randomization
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Started | 174 | 176
Completed | 153 | 159
Not Completed | 21 | 17
Not completed — Death | 1 | 1
Not completed — unresectable | 2 | 3
Not completed — Withdrawal by Subject | 17 | 13
Not completed — Physician Decision | 1 | 0
Period: Surgery
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Started | 153 | 159
Completed (wrong procedure due to screen failure (n=2), failure to notify surgeon of randomization (n=2).) | 152 | 150 (advanced disease=2, inadequate visualization=1, inability to tolerate position=1, colonic mass=1.)
Not Completed | 1 | 9
Not completed — underwent open cystectomy | 0 | 4
Not completed — converted to open procedure | 0 | 5
Not completed — underwent robotic cystectomy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data analysis completed for participants who finished the study as per protocol.
Groups:
- Open Cystectomy: Standard of care treatment, open cystectomy
- Robotic Assisted Radical Cystectomy: Standard of care treatment, robotic assisted radical cystectomy
- Total: Total of all reporting groups
Arm/Group | Open Cystectomy | Robotic Assisted Radical Cystectomy | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Median (Full Range); unit: years] | 67 [37 to 85] | 70 [43 to 90] | 68 [37 to 90]
Sex: Female, Male [Count of Participants; unit: Participants] — Data analysis completed for participants who finished the study as per protocol. Population: Data analysis completed for participants who finished the study as per protocol.
  Participants
    Female | 24 | 24 | 48
    Male | 128 | 126 | 254
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data analysis were completed only for the participants that completed the study.
  Participants
    Hispanic or Latino | 11 | 12 | 23
    Not Hispanic or Latino | 138 | 135 | 273
    Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data analysis completed for participants who finished the study as per protocol. Population: Data analysis completed for participants who finished the study as per protocol.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 10 | 16
    White | 142 | 133 | 275
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 2-year Progression Free Survival (PFS)
Description: Progression will be determined by the treating physician using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria based on radiographic or pathological evidence of disease progression or death from disease.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: percentage of participants
Groups:
- Robotic Assisted Radical Cystectomy: Standard of care treatment using the DaVinci robot.
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
percentage of participants | 71.6 [63.6 to 78.2] | 72.3 [64.3 to 78.8]

2. Primary Outcome: Number of Participants With Positive Margins
Description: Evaluated are the number of participants with positive surgical, bladder, and urethral margins. Positive margin is defined as presence of tumor cells at the edge of the dissected tissue.
Time Frame: At time of cystectomy, approximately 1 hour.
Measure: Count of Participants; unit: Participants
Groups:
- Open Radical Cystectomy: Standard of care treatment, open cystectomy
- Robotic Assisted Radical Cystectomy: Standard of care treatment, robotic assisted radical cystectomy using the DaVinci robot
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
Participants
  Positive surgical margins | 7 | 9
  Positive bladder margins | 5 | 6
  Positive urethral margin | 4 | 3

3. Primary Outcome: Number of Participants Requiring Lymph Node Dissection
Description: Evaluated are the number of participants requiring extended or standard lymph node dissection
Time Frame: At time of cystectomy, approximately 1 hour
Population: 1 participant in the RARC group did not have lymph node dissection.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 149
Participants
  Extended Lymph Node Dissection | 84 | 76
  Standard Lymph Node Dissection | 68 | 73

4. Primary Outcome: Quality of Life (QOL) Outcomes
Description: Functional Assessment of Cancer Therapy- Vanderbilt Cystectomy Index (FACT-VCI) scores range is 0-168 which is sum of physical, emotional, wellbeing, and FACTS Bl Cys. higher scores=better QOL.
Time Frame: at baseline, 3 month, and 6 months
Population: Not all enrolled participants completed the QOL questionnaires.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 111 | 108
score on a scale
  Baseline Visit | 120.9 [115 to 126.8] | 120.1 [114.5 to 125.8]
  3 Month Visit: number analyzed (Participants) | 94 | 97
  3 Month Visit | 125.2 [119.3 to 131.1] | 122.8 [117.2 to 128.3]
  6 Month Visit: number analyzed (Participants) | 91 | 95
  6 Month Visit | 127.5 [121.7 to 133.3] | 126.0 [120.4 to 131.6]

5. Primary Outcome: Number of Participants With Post-surgical Complications
Description: Post surgical complications will be evaluated using the Clavien grading system with scores ranging from 0-5 with the higher number indicating increased post-surgical complications.
Time Frame: 90 days post operative
Population: 90 day complication using Clavien Grading system
Measure: Count of Participants; unit: Participants
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
Participants
  Clavien grade 0 | 47 | 49
  Clavien grade I | 20 | 24
  Clavien grade II | 51 | 44
  Clavien grade III | 28 | 29
  Clavien grade IV | 2 | 0
  Clavien grade V | 4 | 4

6. Primary Outcome: Amount of Estimated Blood Loss (EBL) in ml
Description: Perioperative measures such as EBL will be evaluated by measuring the amount of participant blood loss in ml.
Time Frame: At time of cystectomy, approximately 1 hour
Population: EBL data was not available on 3 of the open radical cystectomy and 2 of the RARC participants.
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 149 | 148
ml | 700 [500 to 1000] | 300 [200 to 500]

7. Primary Outcome: Number of Participants Requiring Blood Transfusion
Description: Number of participants requiring peri, intra, and post operative blood transfusion.
Time Frame: At time of cystectomy, approximately 1 hour
Population: Not all participants in the study required blood transfusion and not all blood transfusion data was available.
Measure: Count of Participants; unit: Participants
Groups:
- Robotic Assisted Radical Cystectomy: Standard of care treatment, robotic assisted radical cystectomy using DaVinci robot
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 143 | 143
Participants
  Perioperative transfusion | 65 | 35
  Intraoperative transfusion: number analyzed (Participants) | 136 | 139
  Intraoperative transfusion | 46 | 18
  Postoperative transfusion: number analyzed (Participants) | 135 | 132
  Postoperative transfusion | 54 | 33

8. Primary Outcome: Number of Days of Post Operative Length of Hospital Stay
Description: Number of days of post operative length of hospital stay will be evaluated
Time Frame: Day 10 post surgery
Population: Not all length of stay data is available for all the study participants.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 146 | 139
days | 7 [6 to 10] | 6 [5 to 10]

9. Primary Outcome: Length of Operative Time
Description: Length of minutes of cystectomy procedure
Time Frame: At time of cystectomy, approximately 1 hour
Population: The length of operative time is not available for all participants.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 146 | 139
minutes | 361 [281 to 450] | 428 [322 to 509]

10. Primary Outcome: Laboratory Values
Description: Serum Hemoglobin (Hb) and Albumin will be reported in grams per deciliters (g/dL)
Time Frame: baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 36 months
Population: Number of participants included was based on the data available at specific time points.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
g/dL
  Baseline (Hb): number analyzed (Participants) | 150 | 148
  Baseline (Hb) | 12.84 (1.87) | 13.11 (1.84)
  6-weeks (Hb): number analyzed (Participants) | 118 | 110
  6-weeks (Hb) | 11.19 (1.58) | 11.62 (1.72)
  3-months (Hb): number analyzed (Participants) | 112 | 108
  3-months (Hb) | 12.05 (1.81) | 12.17 (2.06)
  6-months (Hb): number analyzed (Participants) | 97 | 105
  6-months (Hb) | 12.73 (2.06) | 12.54 (1.89)
  12-months (Hb): number analyzed (Participants) | 81 | 87
  12-months (Hb) | 12.95 (2.48) | 13.25 (2.11)
  24-months (Hb): number analyzed (Participants) | 68 | 73
  24-months (Hb) | 13.47 (1.89) | 13.65 (2.03)
  36-months (Hb): number analyzed (Participants) | 52 | 50
  36-months (Hb) | 14.14 (1.52) | 13.64 (2.59)
  Baseline (Albumin): number analyzed (Participants) | 117 | 123
  Baseline (Albumin) | 3.97 (0.71) | 4.00 (0.55)
  6-weeks (Albumin): number analyzed (Participants) | 98 | 88
  6-weeks (Albumin) | 3.66 (0.62) | 3.70 (0.62)
  3-months (Albumin): number analyzed (Participants) | 97 | 90
  3-months (Albumin) | 3.88 (0.59) | 3.92 (0.60)
  6-months (Albumin): number analyzed (Participants) | 90 | 91
  6-months (Albumin) | 4.02 (0.43) | 4.04 (0.40)
  12-months (Albumin): number analyzed (Participants) | 65 | 75
  12-months (Albumin) | 3.96 (0.93) | 4.04 (0.46)
  24-months (Albumin): number analyzed (Participants) | 58 | 66
  24-months (Albumin) | 4.00 (0.46) | 3.91 (0.75)
  36-months (Albumin): number analyzed (Participants) | 44 | 42
  36-months (Albumin) | 4.00 (0.44) | 3.97 (0.65)

11. Primary Outcome: Measures of Functional Independence as Assessed by the Activities of Daily Living (ADL) Questionnaire
Description: Participant reported ADL questionnaire is a 7 item questionnaire with scores ranging from 7-21 with a lower score indicating increased independence.
Time Frame: baseline, 1 month , 3 months, 6 months
Population: Number of participants changes depending on their data availability at different time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Open Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
score on a scale
  Baseline: number analyzed (Participants) | 138 | 133
  Baseline | 7.2 [7.1 to 7.3] | 7.2 [7.0 to 7.4]
  1-month: number analyzed (Participants) | 125 | 123
  1-month | 7.8 [7.5 to 8.2] | 7.6 [7.3 to 7.9]
  3-months: number analyzed (Participants) | 105 | 109
  3-months | 7.5 [7.1 to 7.8] | 7.3 [7.1 to 7.6]
  6-months: number analyzed (Participants) | 103 | 103
  6-months | 7.1 [7.0 to 7.2] | 7.2 [7.0 to 7.4]

12. Primary Outcome: Percentage of Participants With 3-year Progression Free Survival (PFS)
Description: Progression will be determined by the treating physician using the RECIST Version 1.1 criteria based on radiographic or pathological evidence of disease progression or death from disease.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Open Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
Percent of participants | 65.4 [56.8 to 72.7] | 68.4 [60.1 to 75.3]

13. Primary Outcome: Quality of Life (QOL) Outcomes as Assessed by the Short Form 8 (SF-8) Questionnaire
Description: The SF-8 consists of two component summary scores; physical (PCS) and mental component summary (MCS). They are scored by weighting each score to a norm-based scoring model. The total scores will be reported as a percentile with higher score indicating better quality of health.
Time Frame: baseline, 3 month, and 6 month
Population: Number of participants changes depending on their data availability at different time points.
Measure: Mean (95% Confidence Interval); unit: percentile
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
percentile
  Baseline (PCS): number analyzed (Participants) | 109 | 107
  Baseline (PCS) | 45.3 [43.2 to 47.4] | 46.1 [44.1 to 48.0]
  3-months (PCS): number analyzed (Participants) | 86 | 93
  3-months (PCS) | 46.2 [43.8 to 48.5] | 45.7 [43.5 to 47.9]
  6-months(PCS): number analyzed (Participants) | 93 | 85
  6-months(PCS) | 49.6 [47.6 to 51.7] | 47.5 [45.6 to 49.3]
  Baseline (MCS): number analyzed (Participants) | 109 | 107
  Baseline (MCS) | 48.1 [46.1 to 50.0] | 48.1 [46.4 to 49.9]
  3-months (MCS): number analyzed (Participants) | 86 | 93
  3-months (MCS) | 50.3 [48.6 to 51.9] | 49.1 [47.2 to 51.1]
  6-months(MCS): number analyzed (Participants) | 93 | 85
  6-months(MCS) | 51.8 [50.1 to 53.5] | 49.2 [47.2 to 51.3]

14. Primary Outcome: Total Number of Participants Requiring Intra-operative Fluid Requirement
Description: Total number of participants requiring Intra-operative fluid requirement. (blood+plasma+platelets) Note: In robotic group 1 participant received both plasma and platelets and 1 other received platelets in addition to blood transfusion. In the open group 5 participants received plasma in addition to blood transfusion.
Time Frame: At time of cystectomy, approximately 1 hour
Population: Number of participants included was based on the data available at specific time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 136 | 139
Participants | 46 | 18

15. Primary Outcome: Total Postoperative Analgesic Requirements
Description: Total postoperative analgesic requirements in milli grams
Time Frame: At time of cystectomy, approximately 1 hour
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
mg | 157.7 (222.2) | 167.2 (264.6)

16. Primary Outcome: Creatinine Value.
Description: Serum creatinine will be reported in milligrams per deciliters (mg/dL).
Time Frame: baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 36 months
Population: Number of participants included was based on the data available at specific time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
mg/dL
  Baseline: number analyzed (Participants) | 147 | 148
  Baseline | 1.17 (0.52) | 1.12 (0.50)
  6-weeks: number analyzed (Participants) | 123 | 114
  6-weeks | 1.27 (0.67) | 1.28 (0.66)
  3-months: number analyzed (Participants) | 118 | 110
  3-months | 1.16 (0.44) | 1.26 (0.71)
  6-months: number analyzed (Participants) | 99 | 106
  6-months | 1.21 (0.46) | 1.28 (0.57)
  12-months: number analyzed (Participants) | 82 | 91
  12-months | 1.19 (0.43) | 1.25 (0.58)
  24-months: number analyzed (Participants) | 77 | 82
  24-months | 1.26 (0.48) | 1.25 (0.62)
  36-months: number analyzed (Participants) | 53 | 63
  36-months | 1.26 (0.53) | 1.21 (0.71)

17. Primary Outcome: Measures of Functional Independence as Assessed by the Instrumental Activities of Daily Living (IADL) Questionnaire
Description: Participant reported IADL questionnaire is an 8 item questionnaire with scores ranging from 8-32 with a lower score indicating increased independence.
Time Frame: baseline, 1 month, 3 months, 6 months
Population: Number of participants included was based on the data available at specific time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
score on a scale
  Baseline: number analyzed (Participants) | 136 | 132
  Baseline | 8.8 [8.4 to 9.2] | 8.5 [8.2 to 8.7]
  1-month: number analyzed (Participants) | 122 | 120
  1-month | 10.8 [10.1 to 11.6] | 10.3 [9.6 to 10.9]
  3-months: number analyzed (Participants) | 104 | 105
  3-months | 9.5 [8.8 to 10.1] | 8.9 [8.5 to 9.4]
  6-months: number analyzed (Participants) | 102 | 101
  6-months | 8.6 [8.3 to 9.0] | 8.7 [8.2 to 9.1]

18. Primary Outcome: Performance Related Measures of Functional Independence as Assessed by the Hand Grip Strength Test
Description: The hand grip strength test is measured in kilograms of pressure using a handheld dynamometer.
Time Frame: baseline, 1 month, 3 months, 6 months
Population: Number of participants included was based on the data available at specific time points.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
kg
  Baseline: number analyzed (Participants) | 132 | 127
  Baseline | 37.4 [35.3 to 39.5] | 36.2 [34.3 to 38.2]
  1-month: number analyzed (Participants) | 112 | 104
  1-month | 34.5 [32.4 to 36.6] | 34.1 [31.9 to 36.3]
  3-months: number analyzed (Participants) | 88 | 90
  3-months | 35.1 [32.8 to 37.3] | 34.2 [31.7 to 36.7]
  6-months: number analyzed (Participants) | 86 | 86
  6-months | 36.4 [33.7 to 39.1] | 34.9 [32.3 to 37.5]

19. Primary Outcome: Performance Related Measures of Functional Independence as Assessed by the Time Up and Go (TUG) Walking Test
Description: The TUG test is measured in seconds. Patients will be timed as they rise from a standard chair, walk 3 meters, turn, walk back, and sit again.
Time Frame: baseline, 1 month, 3 months, 6 months
Population: Number of participants included was based on the data available at specific time points.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 152 | 150
seconds
  Baseline: number analyzed (Participants) | 125 | 122
  Baseline | 12.5 [11.2 to 13.7] | 11.7 [10.9 to 12.4]
  1-month: number analyzed (Participants) | 102 | 96
  1-month | 13.6 [12.5 to 14.6] | 13.1 [11.9 to 14.4]
  3-months: number analyzed (Participants) | 83 | 83
  3-months | 12.8 [11.5 to 14.1] | 11.2 [10.5 to 12.0]
  6-months: number analyzed (Participants) | 81 | 81
  6-months | 12.2 [10.6 to 13.8] | 11.2 [10.3 to 12.1]

20. Primary Outcome: Quality of Life (QOL) Outcomes as Assessed by the Functional Assessment of Cancer Therapy - Vanderbilt Cystectomy Index (FACT-VCI) Questionnaire
Description: FACT-VCI consists of eight domains: Five subscale scores (physical wellbeing, social wellbeing, emotional wellbeing, functional wellbeing, and FACT for patients with Bladder Cancer following Cystectomy [FACT-BL-Cys]) and three derived scores (trial outcome index), FACT-General form (FACT-G), and FACT-BL-Cys Total.The ranges of scores for each domain are as follows: 0-28 for physical, social, and functional wellbeing; 0-24 for emotional wellbeing; 0-60 for FACT-BL-Cys; 0-116 for FACT-VCI Trial Outcome Index (sum of physical wellbeing, functional wellbeing, and FACT-BL-Cys scores); 0-108 for FACT-G (sum of physical, social, emotional, and functional wellbeing scores); and 0-168 for FACT-BL-Cys Total (sum of physical, social, emotional, and functional wellbeing scores, and FACT-BL-Cys).The higher score indicates increased wellbeing.
Time Frame: baseline, 3 months, 6 months
Population: Not all participants completed the questionnaire at the different visits.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 115 | 116
score on a scale
  Physical Wellbeing baseline | 23.4 [22.3 to 24.6] | 22.9 [21.8 to 24.0]
  Physical Wellbeing 3 months: number analyzed (Participants) | 102 | 104
  Physical Wellbeing 3 months | 22.8 [21.6 to 24.0] | 23.2 [22.1 to 24.3]
  Physical Wellbeing 6 months: number analyzed (Participants) | 99 | 99
  Physical Wellbeing 6 months | 23.9 [22.7 to 25.0] | 23.2 [22.0 to 24.3]
  Social Wellbeing baseline: number analyzed (Participants) | 115 | 113
  Social Wellbeing baseline | 23.5 [22.2 to 24.8] | 23.5 [22.2 to 24.7]
  Social Wellbeing 3 months: number analyzed (Participants) | 100 | 105
  Social Wellbeing 3 months | 22.6 [21.3 to 23.9] | 23.1 [21.9 to 24.3]
  Social Wellbeing 6 months: number analyzed (Participants) | 98 | 99
  Social Wellbeing 6 months | 23.3 [22.1 to 24.6] | 23.3 [22.1 to 24.5]
  Emotional Wellbeing baseline: number analyzed (Participants) | 112 | 111
  Emotional Wellbeing baseline | 17.7 [16.5 to 18.8] | 17.5 [16.4 to 18.6]
  Emotional Wellbeing 3 months: number analyzed (Participants) | 95 | 98
  Emotional Wellbeing 3 months | 19.9 [18.8 to 21.0] | 19.5 [18.4 to 20.5]
  Emotional Wellbeing 6 months: number analyzed (Participants) | 91 | 96
  Emotional Wellbeing 6 months | 20.0 [18.9 to 21.2] | 19.4 [18.3 to 20.5]
  Functional Wellbeing baseline: number analyzed (Participants) | 115 | 115
  Functional Wellbeing baseline | 18.4 [16.7 to 20.1] | 18.4 [16.8 to 20.0]
  Functional Wellbeing 3 months: number analyzed (Participants) | 100 | 105
  Functional Wellbeing 3 months | 19.3 [17.6 to 21.0] | 17.9 [16.3 to 19.5]
  Functional Wellbeing 6 months: number analyzed (Participants) | 97 | 98
  Functional Wellbeing 6 months | 19.7 [18.0 to 21.4] | 18.5 [16.9 to 20.1]
  FACT-BL-Cys Baseline: number analyzed (Participants) | 114 | 115
  FACT-BL-Cys Baseline | 36.7 [34.2 to 39.2] | 37.4 [35.0 to 39.8]
  FACT-BL-Cys 3 months: number analyzed (Participants) | 100 | 105
  FACT-BL-Cys 3 months | 38.2 [36.0 to 40.5] | 37.9 [35.8 to 40.0]
  FACT-BL-Cys 6 months: number analyzed (Participants) | 97 | 98
  FACT-BL-Cys 6 months | 39.4 [37.1 to 41.6] | 39.3 [37.1 to 41.4]
  Trial outcome index Baseline: number analyzed (Participants) | 114 | 115
  Trial outcome index Baseline | 78.9 [74.3 to 83.5] | 78.9 [74.6 to 83.2]
  Trial outcome index 3 months: number analyzed (Participants) | 100 | 104
  Trial outcome index 3 months | 80.7 [76.3 to 85.2] | 79.3 [75.1 to 83.4]
  Trial outcome index 6 months: number analyzed (Participants) | 97 | 98
  Trial outcome index 6 months | 83.2 [78.8 to 87.6] | 81.1 [77.0 to 85.3]
  FACT-G baseline: number analyzed (Participants) | 112 | 108
  FACT-G baseline | 83.5 [79.5 to 87.4] | 82.4 [78.6 to 86.1]
  FACT-G 3 months: number analyzed (Participants) | 94 | 97
  FACT-G 3 months | 85.8 [81.8 to 89.9] | 84.2 [80.4 to 88.1]
  FACT-G 6 months: number analyzed (Participants) | 91 | 95
  FACT-G 6 months | 87.4 [83.5 to 91.4] | 85.9 [82.1 to 89.7]
  FACT-BL-Cys Total baseline: number analyzed (Participants) | 111 | 108
  FACT-BL-Cys Total baseline | 120.9 [115.0 to 126.8] | 120.1 [114.5 to 125.8]
  FACT-BL-Cys Total 3 months: number analyzed (Participants) | 94 | 97
  FACT-BL-Cys Total 3 months | 125.2 [119.3 to 131.1] | 122.8 [117.2 to 128.3]
  FACT-BL-Cys Total 6 months: number analyzed (Participants) | 91 | 95
  FACT-BL-Cys Total 6 months | 127.5 [121.7 to 133.3] | 126.0 [120.4 to 131.6]

21. Secondary Outcome: Cost
Description: Fixed and variable costs associated with the procedure.
Time Frame: Day 7
Population: Cost data was specified as a secondary endpoint in the protocol, but data could not be collected from all sites due to proprietary reasons.
Arm/Group | Open Radical Cystectomy | Robotic Assisted Radical Cystectomy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 month
Description: Adverse events (AE) are defined as complications related to the robotic/open cystectomy and/or study procedures as determined by the principal investigator.
Arm/Group | Open Cystectomy | Robotic Assisted Radical Cystectomy
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/150
Other Adverse Events (participants affected / at risk) | 105/152 | 101/150
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Cystectomy (N=152) | Robotic Assisted Radical Cystectomy (N=150)
Urinary Tract Infection (Renal and urinary disorders) | 39 (39) | 53 (53)
post operative ileaus (Gastrointestinal disorders) | 31 (31) | 33 (33)
Anastomotic bowel leak (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 6 (6) | 6 (6)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 4 (4)
Sepsis (Infections and infestations) | 16 (16) | 15 (15)
Superficial wound infection (Infections and infestations) | 18 (18) | 11 (11)
Deep wound infection (Infections and infestations) | 10 (10) | 3 (3)
Intra-abdominal infection (Infections and infestations) | 3 (3) | 7 (7)
Stoma site infection (Infections and infestations) | 3 (3) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 19 (19) | 17 (17)
Renal insufficiency requiring dialysis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Fistula (Renal and urinary disorders) | 2 (2) | 3 (3)
Ureteral Stricture (Renal and urinary disorders) | 10 (10) | 13 (13)
Intestinal stoma leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Ureteric anastomotic leak (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Wound disruption (Injury, poisoning and procedural complications) | 11 (11) | 7 (7)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Failure to wean from vent within 48 hours of surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Re-intubation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lymphocele (Vascular disorders) | 3 (3) | 4 (4)
Pulmonary embolism (Vascular disorders) | 4 (4) | 4 (4)
Thromboembolic event (Vascular disorders) | 12 (12) | 7 (7)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 7 (7)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac event with cardiopulmonary resuscitation (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT01157676/Prot_SAP_000.pdf